CLINICAL TRIAL: NCT02816554
Title: Safety and Immunogenicity of an Inactivated Japanese Encephalitis Vaccine (JECEVAX) in Vietnamese Children
Brief Title: Safety and Immunogenicity of JECEVAX in Young Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Hygiene and Epidemiology, Vietnam (Other)
Collaborators: Ministry of Science and Technology, Vietnam (Other Government); Ministry of Health, Vietnam (Other Government)
Responsible Party: Principal Investigator, Vu Dinh Thiem, Head, Department of Epidemiology, National Institute of Hygiene and Epidemiology, Vietnam
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2015-JECEVAX-2R
Record Dates: First submitted 2016-06-23; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Japanese Encephalitis
Keywords: Japanese Encephalitis; JECEVAX; Vietnam
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- JECEVAX-1 (Experimental): JECEVAX - VABIOTECH Vietnam Liquid form Composition: 1.0 BR209 Subcutaneous injection 0.5ml/dose, 2 doses, interval 10-12days
  Interventions: Biological: JECEVAX-1
- JECEVAX-0.8 (Experimental): JECEVAX - VABIOTECH Vietnam Liquid form Composition: 0.8 BR209 Subcutaneous injection 0.5ml/dose, 2 doses, interval 10-12 days
  Interventions: Biological: JECEVAX-0.8
- JECEVAX-0.5 (Experimental): JECEVAX - VABIOTECH Vietnam Liquid form Composition: 0.5 BR209 Subcutaneous injection 0.5ml/dose, 2 doses, interval 10-12 days
  Interventions: Biological: JECEVAX-0.5
- JEVAX (Active Comparator): JEVAX - VABIOTECH Vietnam Liquid form Composition: 1,0 BR209 Subcutaneous injection 0.5ml/dose, 2 doses, interval 10-12 days
  Interventions: Biological: JEVAX

INTERVENTIONS:
Biological: JEVAX — JEVAX - VABIOTECH Vietnam Liquid form Subcutaneous injection 0.5ml/dose, 2 doses, 10-12 days interval
  Arms: JEVAX
Biological: JECEVAX-1 — JECEVAX - VABIOTECH Vietnam Liquid form Composition: 1 BR209 Subcutaneous injection 0.5ml/dose, 2 doses, interval 10-12 days
  Other Names: JECEVAX-HI
  Arms: JECEVAX-1
Biological: JECEVAX-0.8 — JECEVAX - VABIOTECH Vietnam Liquid form Composition: 0.8 BR209 Subcutaneous injection 0.5ml/dose, 2 doses, interval 10-12 days
  Other Names: JECVAX-MED
  Arms: JECEVAX-0.8
Biological: JECEVAX-0.5 — JECEVAX - VABIOTECH Vietnam Liquid form Composition: 0.5 BR209 Subcutaneous injection 0.5ml/dose, 2 doses, interval 10-12 days
  Other Names: JECEVAX-LOW
  Arms: JECEVAX-0.5

SUMMARY:
A dose escalating study with 3 different dosing regimens of the studied vaccine (JECEVAX- VABIOTECH-Vietnam) and a licensed vaccine (JEVAX-VABIOTECH-Vietnam) is conducted in Vietnamese children, aged 9 to 24 months to assess the safety and immunogenicity. Two hundred children are enrolled and randomly assigned into 4 groups (50 children/group), each of which receive 2 doses of study / control vaccine subcutaneously, at 10-12 days interval. Safety issues included immediate reaction at the site of injection and systemic reaction within 30 min of administration, solicited and unsolicited adverse events occurs from the first dose to 30 days after second dose; SAE (from start of first dose to 30 days after second dose), blood cell count, urea, ALT, AST. Immunogenicity outcomes include seroconversion of neutralizing antibodies (blood samples are taken prior to 1st dose and 20-22 days post 2nd dose).

DETAILED DESCRIPTION:
Mouse brain-derived Japanese Encephalitis (JE) vaccine was developed in Vietnam since 1989 with the support from WHO and BIKEN institute, Japan. It helped Viet Nam prevents Japanese Encephalitis outbreaks successfully during those years.

However, mouse brain-derived JE vaccine production requires companies to compliance various requirements from WHO. Especially, WHO has a plan to replace the mouse brain-derived JE vaccines with Cell culture-derived JE vaccines.

Vero cell-derived vaccine technology shows many advantages compares to Mouse brain-derived vaccine technology. VABIOTECH has been approved and sponsored by the Ministry of Science and Technology to produce Vero cell - derived JE vaccine. The vaccine demonstrated a good safety and immunogenicity profile in animal models. The vaccine has been proven safety in volunteer adults.

In this study, a dose escalating study with 3 different dosing regimens of the studied vaccine (JECEVAX) and a licensed vaccine (JEVAX-VABIOTECH Vietnam) is conducted in Vietnamese children, aged 9-24 months to assess the safety and immunogenicity. Two hundred children are enrolled and randomly assigned into 4 groups (50 children/group), each of which receive 2 doses of investigate vaccines or control vaccine subcutaneously, at 10-12 days interval. Safety issues included immediate reaction at the site of injection and systemic reaction within 30 min of administration, solicited and unsolicited adverse events occurs from the first dose to 30 days after second dose; SAE (from start of first dose to 30 days after second dose), blood cell count, urea, ALT, AST. Immunogenicity outcomes include seroconversion of neutralizing antibodies (blood samples are taken prior to 1st dose and 20-22 days post 2nd dose).

ELIGIBILITY:
Inclusion Criteria:

* Healthy children of both sexes, 9-24 months of age;
* Have not been vaccinated with JE vaccine;
* Not have any chronic disease;
* Parents/legal guardians agree to participate their children in this study and sign the informed consent.

Exclusion Criteria:

* Currently has chronic diseases (cardiovascular, liver and spleen related etc);
* Currently has acute diseases;
* Use (orally or injection) with corticosteroid containing drug (>1 mg / kg dose);
* Use of immunocompromised treatment within 4 weeks of enrollment;
* Being immunocompromised and autoimmune diseases (HIV, lupus);
* The family history of immunocompromised;
* History of febrile seizure;
* Allergic to any vaccine component;
* Fever (>38 Celsius degree) within 3 days before vaccination or at enrollment;
* Malnourished (3rd grade or above);
* Blood disorder;
* Use of vaccines which have not been licenced 7 days before enrolment in this study

Ages: 9 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events during study period. | Up to 30 days after 2nd dose
  Number of participants with solicited and unsolicited adverse events after each dose of vaccine: immediately injection site and systemic AEs after vaccination (within 30 min), solicited and unsolicited AEs within 7 days after each dose, unsolicited AEs from day 8 after dose 1 to date of dose 2 and from day 8 after dose 2 to day 30 post 2nd dose, as assessed by CTCAE v.4.0.
Number of participants have sero-conversion at 20-22 days post 2nd dose (compared to pre-vaccination) | Up to 20-22 days after the 2nd dose
  Sero-conversion rate of each JECEVAX regimen and JEVAX at 20-22 days after 2 doses of vaccines

SECONDARY OUTCOMES:
Number of participants with treatment-related SAE during study period | Up to 30 days after the 2nd dose
  Number of participants with treatment-related SAE during study period of JECEVAX compared to that of JEVAX, as assessed by CTCAE ver 4.0
Number of participants with abnormal laboratory value. | Up to 20-22 days after the 2nd dose.
  Numbers of participants with abnormal laboratory values (blood cell counts, urea concentration, liver function (ALT, AST concentration) when administered with different JECEVAX formulations and with JEVAX before the first dose and 20-22 days after the 2nd dose.

CONTACTS AND LOCATIONS:
Overall Officials: Thiem D Vu, MD., PhD., Principal Investigator — National Institute of Hygiene and Epidemiology, Vietnam
Locations (2):
- Vietnam (2):
  - District Health Center, Thanh Sơn, Phu Tho
  - Phu Tho Preventive Medicine Center, Việt Trì, Phu Tho

IPD SHARING:
Plan to Share IPD: No
Individual data with identification removed are to be available for Ethical committee, Ministry of Health and National Foundation of Science and Technology Development to avoid misuse of data.
  Public shared data will be in the form of summarised tables and figures.